CLINICAL TRIAL: NCT03268070
Title: Targeting Motor Areas for Customized Transcranial Magnetic Stimulation in Motor Rehabilitation Treatment of Chronic Stroke Patients
Brief Title: Transcranial Magnetic Stimulation in Stroke Motor Rehabilitation Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is withdrawn due to funding.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Cathrin Buetefisch, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00097855
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Transcranial Magnetic Stimulation; Neurophysiology; Neuroscience; Stroke Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinded to the type of TMS that they receive on each day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Repetitive TMS over contralateral premotor cortex (Experimental): Location of repetitive Transcranial Magnetic Stimulation (rTMS): contralateral premotor cortex.
  Interventions: Device: Repetitive TMS over contralateral premotor cortex.
- Repetitive TMS over ipsilateral premotor cortex (Experimental): Location of repetitive Transcranial Magnetic Stimulation (rTMS): ipsilateral premotor cortex.
  Interventions: Device: Repetitive TMS over ipsilateral premotor cortex.
- Repetitive TMS over contralateral primary motor cortex (Experimental): Location of repetitive Transcranial Magnetic Stimulation (rTMS): contralateral primary motor cortex.
  Interventions: Device: Repetitive TMS over contralateral primary motor cortex.
- Sham repetitive TMS over contralateral premotor cortex (Sham Comparator): Location of Sham repetitive Transcranial Magnetic Stimulation (rTMS): contralateral premotor cortex.
  Interventions: Device: Sham Repetitive TMS over contralateral premotor cortex.
- Single TMS over extensor carpi ulnaris spot of motor cortex (Experimental): Location of single-pulse Transcranial Magnetic Stimulation (sTMS): extensor carpi ulnaris (ECU) hotspot of primary motor cortex (M1).
  Interventions: Device: Single TMS over extensor carpi ulnaris spot of motor cortex

INTERVENTIONS:
Device: Repetitive TMS over contralateral premotor cortex. — Repetitive Transcranial magnetic stimulation (rTMS) will be applied over contralateral premotor cortex during motor training. TMS uses magnetism to excite neurons near the surface of the brain. Frequency of rTMS: 0.1 Hz; time of rTMS: 50 milliseconds before the onset of movement-related electromyography (EMG); device: Super Rapid 2 Transcranial Magnetic Stimulator.
  Arms: Repetitive TMS over contralateral premotor cortex
Device: Repetitive TMS over ipsilateral premotor cortex. — Repetitive Transcranial magnetic stimulation (rTMS) will be applied over ipsilateral premotor cortex during motor training. TMS uses magnetism to excite neurons near the surface of the brain. Frequency of rTMS: 0.1 Hz; time of rTMS: 50 milliseconds before the onset of movement-related electromyography (EMG); device: Super Rapid 2 Transcranial Magnetic Stimulator.
  Arms: Repetitive TMS over ipsilateral premotor cortex
Device: Repetitive TMS over contralateral primary motor cortex. — Repetitive Transcranial magnetic stimulation (rTMS) will be applied over contralateral primary motor cortex during motor training. TMS uses magnetism to excite neurons near the surface of the brain.Frequency of rTMS: 0.1 Hz; time of rTMS: 50 milliseconds before the onset of movement-related electromyography (EMG); device: Super Rapid 2 Transcranial Magnetic Stimulator.
  Arms: Repetitive TMS over contralateral primary motor cortex
Device: Sham Repetitive TMS over contralateral premotor cortex. — Sham rTMS will be applied over contralateral premotor cortex. TMS uses magnetism to excite neurons near the surface of the brain. Frequency of rTMS: 0.1 Hz; time of rTMS: 50 milliseconds before the onset of movement-related electromyography (EMG); device: Super Rapid 2 Transcranial Magnetic Stimulator.
  Arms: Sham repetitive TMS over contralateral premotor cortex
Device: Single TMS over extensor carpi ulnaris spot of motor cortex — Single-pulse TMS will be applied over the extensor carpi ulnaris (ECU) hotspot of primary motor cortex (M1) during motor training.TMS uses magnetism to excite neurons near the surface of the brain. TMS pulses will be applied at different strengths (30%-80% maximum stimulator output) and record subsequent activity of the ECU muscle using electromyography (EMG).
  Arms: Single TMS over extensor carpi ulnaris spot of motor cortex

SUMMARY:
The goal of the study is to determine the effect of repetitive transcranial magnetic stimulation (rTMS) over the premotor cortex on training-related improvements in motor performance and associated neural plasticity.

DETAILED DESCRIPTION:
Occlusion of the middle cerebral artery is the most common cause of stroke. Because the middle cerebral artery supplies blood to the motor cortices, middle cerebral artery stroke often impacts the integrity of the motor cortex and its associated corticospinal projections. Less than half of all individuals post-stroke regain complete motor function. Because motor deficits, especially of the upper extremities, can dampen the quality of life, there is an urgent need to improve current rehabilitation programs to allow more stroke survivors to achieve higher functional gains.

Motor training is an important part of recovery after stroke. During motor training, patients practice performing a movement and become better at performing the trained movement over time. Repetitive transcranial magnetic stimulation (rTMS), which uses magnetism to excite neurons near the surface of the brain, may further improve performance. There is evidence that the premotor cortex may be a more effective target than the primary motor cortex for rTMS for some stroke survivors. In the current study, the investigator will determine the effect of rTMS over the premotor cortex on training-related improvements in motor performance in adults who experienced a stroke more than 6 months ago.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to give informed, written consent
* Be aged 30-80 years old
* Have a single ischemic infarction affecting the primary motor system
* Have intact cognitive abilities
* No current depression
* No neurological disease
* No contradictions to TMS

  * No history of seizures or epilepsy
  * No implanted medical device
  * No metal in neck or head
  * No history of migraine headaches
  * No intake of medication that lowers seizure threshold

Exclusion Criteria:

* none

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in wrist velocity | Before, 0 mins after, 30 mins after, and 60 mins after motor training.
  The subjects will be asked to perform 7 isometric wrist extensions before and after motor training. Wrist velocity will be measured by a gyroscope taped to the dorsum of the wrist that was used during motor training. An increase in the maximum velocity that persists at least an hour after training is indicative of motor learning.
Change in Stimulus Response Curve parameters | Before, 0 mins after, 30 mins after and 60 mins after motor training.
  To measure organization of a motor region in the primary motor cortex supporting wrist movement, a Stimulus Response Curve (SRC) will be collected before and after motor training. SRC is a set of motor evoked potentials (MEP) that characterizes input-output parameters of the primary motor cortex and associated corticospinal tract. A change in the SRC parameters after training will reflect a change in the organization of the primary motor cortex.

SECONDARY OUTCOMES:
Change in wrist force | Before, 0 mins after, 30 mins after, and 60 mins after motor training.
  The subjects will be asked to perform 7 isometric wrist extensions before and after motor training. A force transducer will record the maximum force produced during the wrist extensions.
Change in reaction time | Before, 0 mins after, 30 mins after and 60 mins after motor training.
  Subjects will be asked to perform 7 auditory-cued ballistic wrist extensions before and after motor training. Electromyographic (EMG) activity recorded during the ballistic wrist extensions will be used to measure reaction time. Reaction time is the length of time between the auditory cue and the onset of the movement-related EMG burst of the extensor carpi ulnaris muscle.
Change in task accuracy | During motor training (will compare first block to last block).
  Task accuracy will be determined by the number of successful trials over the number of total trials. A trial will be considered successful when the subject moves a cursor from the home position into a target box by modulating the acceleration of their wrist. An increase in task accuracy after training will indicate motor learning.
Change in Short interval intracortical inhibition (SICI) of the primary motor cortex | Before, 0 mins after, 30 mins after, and 60 mins after motor training.
  Short interval intracortical inhibition (SICI) is an inhibitory phenomenon in the motor cortex. To test for SICI, a sub-threshold conditioning stimulus (CS) will precede a supra-threshold test stimulus (TS) by 2 milliseconds. The amplitude of a conditioned TS-evoked MEP will be expressed as a percent of the amplitude of an unconditioned TS-evoked MEP (% MEP). A decrease in the % MEP after training would indicate a increase in SICI. An increase in the % MEP after training would indicate a decrease in SICI.
Change in Resting Motor Threshold | Before, 0 mins after, 30 mins after, and 60 mins after motor training.
  Parametric Estimation by Sequential Testing (PEST) will be used to determine the Resting Motor Threshold (rMT). The mathematical algorithm implemented by PEST will determine the rMT with fewer TMS pulses than the traditional method.

CONTACTS AND LOCATIONS:
Overall Officials: Cathrin Buetefisch, MD, Principal Investigator — Emory University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available for sharing with other researchers. Data will be shared with the Enhancing Neuroimaging Genetics through Meta-Analysis (ENIGMA) Stroke Recovery group. The researchers plan to share the entire data set including clinical, behavioral, anatomical MRI data, with the ENIGMA Stroke Recovery group.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data will be available for sharing following publication of primary results from this study, with no end date for sharing.
Access Criteria: The format of the shared data will be compatible with the ENIGMA data base. Outside researchers interested in using this data can contact Dr. Buetefisch at cathrin.buetefisch@emory.edu.